CLINICAL TRIAL: NCT05459831
Title: Efficacy Comparison of High and Very High Power Short Duration Pulmonary Vein Isolation
Acronym: HPSD-Remap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Nandor Szegedi, Assistant Professor, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BWI- IIS-653
Record Dates: First submitted 2022-07-04; First posted 2022-07-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; high-power, short-duration; pulmonary vein isolation; durability
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary vein isolation with 50W energy setting (Active Comparator): In this group of subjects, the initial pulmonary vein isolation procedure will be performed using 50W radiofrequency energy. This power setting will be used for all the ablation points.
  Interventions: Device: QDot Micro Catheter
- Pulmonary vein isolation with 90W energy setting (Active Comparator): In this group of subjects, the initial pulmonary vein isolation procedure will be performed using 90W radiofrequency energy. This power setting will be used for all the ablation points.
  Interventions: Device: QDot Micro Catheter

INTERVENTIONS:
Device: QDot Micro Catheter — Atrial fibrillation radiofrequency ablation with 90W or 50W energy setting.

SUMMARY:
Objective: To evaluate the long-term durability of PVI performed with 90W and 50W (QDot catheter).

Primary hypothesis: Pulmonary vein isolation performed with 90W (QMODE+) and inter-tag distance <5 mm is non-inferior to pulmonary vein isolation performed with 50W guided by ablation index (QMODE) and inter-tag distance <5 mm.

Study Design: 40 patients will be randomized in a 1:1 ratio to 50W and 90W PVI.

Study procedures: Initial PVI will be performed via femoral access and double transseptal puncture guided by fluoroscopy and pressure monitoring. If necessary intracardiac echocardiography (ICE) will be used for the transseptal puncture. A fast anatomical left atrial map will be created with a multipolar mapping catheter; then, point-by-point PVI will be performed with QDot catheter with 50W or 90W according to randomization. Three months after the initial procedure, patients will undergo a repeated high density left atrial mapping with PentaRay or OctaRay catheter to evaluate the durability of the PVI. Exact gap numbers and locations will be registered. If necessary, reablation of the pulmonary veins (rePVI) will be performed.

Inclusion criteria: Symptomatic paroxysmal/persistent AF, >18 years, willingness to sign informed consent form.

Exclusion criteria: Long-standing persistent AF, active malignancy, contraindication for anticoagulant therapy, life expectancy <1 year, valvular AF, hyperthyroidism.

Endpoints: At repeat procedure, a high density left atrial map will be created with PentaRay or if available OctaRay catheter to evaluate the durability of the PVI. Primary endpoint will be pulmonary vein reconnection.

DETAILED DESCRIPTION:
1. Background

   Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia in adults. Its prevalence increases with age, affecting 3/100 people, and its incidence is also correlated with age, affecting 30/100,000 people per year. Its clinical significance stems from common complications (stroke, heart failure) and concomitant higher mortality.

   The most effective treatment method of atrial fibrillation is catheter ablation, which seeks to maintain sinus rhythm. Isolation of the triggering pulmonary veins (PVI) from the left atrium is the cornerstone of AF ablation. PVI has undergone significant technical development over the past decade; however, the chances of arrhythmia recurrence and the occurrence of procedural complications are not negligible.

   Experiments have shown that lesions with a larger surface diameter but less depth develop during HPSD ablation; the higher the energy is, the shallower and wider the lesions are. These lesion properties make it easier to create a solid line from the ablation points, while the shallower lesion causes less damage to the surrounding tissues. The latest application of HPSD technology is the so-called "very high power short duration" (vHPSD) ablation when we apply 90W power. No data are available on long-term efficacy or safety comparing ablation with HPSD vs. vHPSD.
2. Objective: To evaluate the durability of radiofrequency PVI performed with 90W (QMODE plus) and 50W (QMODE) with the QDot catheter.
3. Primary hypothesis: Pulmonary vein isolation performed with 90W (QMODE+) and inter-tag distance <5 mm is non-inferior to pulmonary vein isolation performed with 50W guided by ablation index (QMODE) and inter-tag distance <5 mm.
4. Study Design: Single-center, prospective, randomized study. Patients will be randomly assigned in a 1:1 ratio to HPSD (50W) and vHPSD (90W) PVI.
5. Research period Planned research period from the second quarter of 2022 for a maximum of 1 year.
6. Study subjects

   • Planned number of included subjects: 40.
7. Study procedures:

   * Initial PVI will be performed via femoral access after double transseptal puncture guided by fluoroscopy and pressure monitoring. If necessary ICE will be used for the transseptal puncture. A fast anatomical left atrial map will be created with a multipolar mapping catheter; then, point-by-point PVI will be performed with QDot catheter with 50W or 90W according to randomization. After creating the isolation circle, the presence or absence of first-pass isolation will be assessed by multipolar catheters. If PVI is not complete at this point, it will be completed to reach complete isolation of all veins. After that, a 20 minutes waiting period will be the next step to evaluate presence or absence of acute reconnection of the PV-s. In case of acute reconnection, touch-up applications will be delivered to complete the PVI.
   * Three months after the initial procedure, patients will undergo a repeated high density left atrial mapping with PentaRay or, if available OctaRay catheter to evaluate the durability of the PVI. Exact gap numbers and locations will be registered (based on the 16 segment PV model). If necessary, rePVI will be performed.
8. Statistical analysis Continuous variables are expressed as mean and standard deviation, or median and interquartile ranges, depending on the normal of non-normal distribution. Categorical variables are expressed in numbers and percentages. Continuous variables are compared by parametric or non-parametric tests, depending on the distribution, while categorical variables are compared by Chi-square test or Fisher's exact test. The predictive value of different ablation techniques in outcome is planned to be analyzed by logistic regression. A two-tailed p-value of <0.05 will be considered statistically significant. Statistical analyses will be performed using IBM SPSS 25 (Apache Software Foundation, USA) and GraphPad Prism 7.1 (GraphPad Softwares Inc., USA) software products.
9. Data management All study patient data is entered into Semmelweis University's electronic database (accessible only from Semmelweis University's network) in a coded and unique manner, with a unique identifier, to which project staff has a password-protected, defined level of access. Each person involved in the study is given a unique identification code, and the data stored in the database is linked to that unique identifier. Thus, a data set will be incomprehensible and unusable for an external (unauthorized) user. The data belonging to the unique identification code, with which the patient's identity can be clearly indicated (name, place and date of birth, clinical reference number, identification number, identity card number, etc.) are not available from the database and are stored separately from it. Access to personal data is restricted to institutional leaders and program professional leaders.
10. Personal and material requirements The personal and material requirements of the research are available at the Heart and Vascular Center of Semmelweis University. The personal requirements are given by the staff of the Electrophysiological Laboratory, and the material conditions are provided by the equipment of the same laboratory.
11. Ethics approval

An ethics approval was obtained from the Hungarian National Public Health Center (No. 8119-2/2022/EÜIG).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal/persistent AF
* Age >18 years
* Willingness to sign informed consent form.

Exclusion Criteria:

* Contraindication to ablation
* Contraindication of long-term anticoagulation
* Long-standing persistent AF
* History of PVI
* History of cardiac surgery
* Pregnancy
* Active malignancy
* Life expectancy <1 year
* Valvular AF
* Reversible cause of AF (e.g. hyperthyroidism).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary vein reconnection | 3 month
  Presence or absence of pulmonary vein reconnection at 3 month remapping procedure

SECONDARY OUTCOMES:
Procedure time | Immediately after the procedure
  Procedure time of the initial pulmonary vein isolation procedure
Fluoroscopy time | Immediately after the procedure
  Fluoroscopy time of the initial pulmonary vein isolation procedure
Fluoroscopy dose | Immediately after the procedure
  Fluoroscopy dose of the initial pulmonary vein isolation procedure
Major complication | 3 month
  Major complication of the initial pulmonary vein isolation procedure
First pass isolation | Immediately after the procedure
  First pass isolation during the initial pulmonary vein isolation procedure
Acute reconnection | Immediately after the procedure
  Acute reconnection during the initial pulmonary vein isolation procedure
Major complication of the second (remapping) procedure | 1 week
  Major complication of the second (remapping) procedure
12-month atrial fibrillation freedom | 12 months
  freedom from atrial fibrillation during the 12-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: László Gellér, Ph.D., DSc, Study Chair — Semmelweis University
Locations (1):
- Semmelweis University, Budapest, Hungary

REFERENCES:
- [Derived] Szegedi N, Sallo Z, Nagy VK, Osztheimer I, Hizoh I, Lakatos B, Boussoussou M, Orban G, Boga M, Ferencz AB, Komlosi F, Toth P, Perge P, Kovacs A, Merkely B, Geller L. Long-Term Durability of High- and Very High-Power Short-Duration PVI by Invasive Remapping: The HPSD Remap Study. Circ Arrhythm Electrophysiol. 2024 Feb;17(2):e012402. doi: 10.1161/CIRCEP.123.012402. Epub 2024 Jan 29. PMID 38284286